CLINICAL TRIAL: NCT05776420
Title: Effect of a Healthy Food Voucher on Blood Glucose Control in People With Type 2 Diabetes or Prediabetes: a Randomized Controlled Trial
Brief Title: Effect of a Healthy Food Voucher on Blood Glucose Control in People With Type 2 Diabetes or Prediabetes
Acronym: VOUCH4DIABETES
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21-112
Record Dates: First submitted 2023-02-03; First posted 2023-03-20 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-02

CONDITIONS: Diabete Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Food voucher (Experimental): $65 monthly voucher for healthy foods (phase 1)
  Interventions: Behavioral: Food voucher
- Control (No Intervention)
- Large voucher (Experimental): $160 monthly voucher for healthy foods (phase 2)
  Interventions: Behavioral: Food voucher
- Small voucher (Active Comparator): $40 monthly voucher for healthy foods (phase 2)
  Interventions: Behavioral: Food voucher

INTERVENTIONS:
Behavioral: Food voucher — A voucher of that can be redeemed for food at grocery stores.
  Arms: Food voucher; Large voucher; Small voucher

SUMMARY:
This randomized controlled trial (RCT) will determine if access to a voucher for healthy foods reduces blood sugar levels among people living on a low income who have type 2 diabetes or elevated blood sugar.

ELIGIBILITY:
Inclusion Criteria:

* hemoglobin A1c 6.0 to 11.0
* report food insecurity or financial insecurity

Exclusion Criteria:

* live with a current study participant
* life expectancy < 6 months
* multiple life-threatening allergies to common foods
* require total parenteral nutrion
* blood dyscrasia that interferes with hemoglobin A1c interpretation
* hemoglobin A1c >11

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1c | 6 months
  Change in hemoglobin A1c

SECONDARY OUTCOMES:
General health ("In general, how would you rate your health today?") | 6 months
  Self-reported health. Potential responses are: very good, good, moderate, bad, very bad and decline to respond.
Financial security ("Do you have trouble making ends meet at the end of the month?") | 6 months
  Self-reported financial security
Food insecurity measured by 6 questions from Household Food Security Survey | 6 months
  Self-reported food insecurity
Fruit and vegetable consumption | 6 months
  Self-reported fruit and vegetable consumption
Health care utilization using administrative data | 6 months
  Includes hospitalizations, outpatient visits and primary care visits
Carotenoid level | 6 months
  Serum caortenoid level

CONTACTS AND LOCATIONS:
Locations (1):
- St Michael's Hospital Academic Family Health Team, Toronto, Canada

IPD SHARING:
Plan to Share IPD: Yes
We plan to share de-identified individual participant data

REFERENCES:
- [Derived] Persaud N, Ul Haq MZ, Buadu A, Sabir A, Sinha L, Thorpe KE, Xu K, Hwang SW, Pinto AD, Gucciardi E. Voucher for Healthy Foods and Diabetes Control: A Randomized Clinical Trial. JAMA Intern Med. 2025 Dec 1;185(12):1434-1441. doi: 10.1001/jamainternmed.2025.5420. PMID 41114992